CLINICAL TRIAL: NCT00285467
Title: Comparison of Cholecalciferol Versus Doxercalciferol in the Treatment of Secondary Hyperparathyroidism in CKD
Brief Title: Cholecalciferol Versus Doxercalciferol in the Treatment of Secondary Hyperparathyroidism in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0508-06
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Renal Osteodystrophy
Keywords: kidney, parathyroid hormone, vitamin d
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder | interventions — 1 alpha-hydroxyergocalciferol; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxercalciferol (Experimental): doxercalciferol 1 mcg capsule orally daily for 3 months. This is a form of vitamin D that does not require activation by enzymes in the liver and kidney.
  Interventions: Drug: doxercalciferol
- Cholecalciferol (Active Comparator): cholecalciferol 4000 IU capsule orally daily for one month, then 2000 IU capsule daily orally for 2 months. this form of vitamin D requires activation by cells of the body.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: doxercalciferol — form of vitamin D that is already in active form.
  Other Names: Hectoral
  Arms: Doxercalciferol
Drug: Cholecalciferol — from of vitamin D that requires cells in the body to make active
  Other Names: vitamin D3
  Arms: Cholecalciferol

SUMMARY:
The majority of patients with moderate to severe chronic kidney disease (CKD) (stages 3 and 4) develop secondary hyperparathyroidism (2°HPT), but the optimal therapy to control hyperparathyroidism in this group is unknown. The National Kidney Foundation presented guidelines in 2003 recommending vitamin D supplementation for vitamin D insufficient patients and active vitamin D therapy in patients with sufficient levels. These guidelines are based on opinion since there are no significant trials to determine if vitamin D supplementation is effective in this population. The active vitamin D metabolites doxercalciferol, paricalcitol, and calcitriol have been shown to effectively suppress parathyroid hormone (PTH), but have not been compared with vitamin D supplementation with a calciferol (ergocalciferol or cholecalciferol). Beyond hyperparathyroidism, small studies suggest vitamin D replacement in vitamin D insufficient non-CKD subjects result in improved pain, feeling of well being, blood pressure and strength. In this proposed study we wish to directly compare the effectiveness of cholecalciferol versus doxercalciferol in suppressing elevated PTH levels in subjects with CKD not on dialysis who have vitamin D insufficiency in a three month study. Secondary endpoints will be change in blood pressure.

DETAILED DESCRIPTION:
Patients with CKD stage 3 were randomly allocated (by blinded group allocation) to either cholecalciferol (4000 U per day for one month then 2000 IU daily thereafter) or doxercalciferol (2.5 mcg po daily. Assessments for blood endpoints (primary end point PTH; secondary calcium, phosphorus) were done monthly. Other assessments (blood pressure) were done at baseline and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years old or older, male or female
* able to sign informed consent
* CKD stage 3 (GFR 30-59 ml/min) or stage 4 (15-29 ml/min)
* intact Parathyroid hormone level (iPTH) > 100 pg/ml for stage 3 or iPTH > 150 pg/ml for stage 4
* calcidiol levels ≤ 20 ng/ml
* ability to ambulate without assistance

Exclusion Criteria:

* intact PTH > 400 pg/ml
* initial corrected Calcium > 9.7 mg/dl
* initial serum Phosphorous > 5.0 mg/dl
* initial standardized blood pressure of > 160/100
* history of significant liver disease or cirrhosis
* anticipated requirement for dialysis in 6 months
* malabsorption, severe chronic diarrhea, or ileostomy
* no calcimimetic or active vitamin D therapy 30 days prior to enrollment
* use of digoxin, magnesium containing products, mineral oil, or cholestyramine

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Moe, MD, Study Director — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moe SM, Saifullah A, LaClair RE, Usman SA, Yu Z. A randomized trial of cholecalciferol versus doxercalciferol for lowering parathyroid hormone in chronic kidney disease. Clin J Am Soc Nephrol. 2010 Feb;5(2):299-306. doi: 10.2215/CJN.07131009. Epub 2010 Jan 7. PMID 20056760

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxercalciferol, Active Vitamin D: Doxercalciferol is an active Vitamin D readily usable by human body.
- Cholecalciferol, Inactive Vitamin D: Cholecalciferol is inactive Vitamin D and requires the kidneys to make it active.
Period: Overall Study
Arm/Group | Doxercalciferol, Active Vitamin D | Cholecalciferol, Inactive Vitamin D
Started | 25 | 22
Completed | 25 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 47 subjects had at least one follow up visit after taking medications and were included in results.
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxercalciferol, Active Vitamin D | Cholecalciferol, Inactive Vitamin D | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 62 (10) | 63.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants] — 55 subjects were consents and underwent qualifying blood tests. 47 subjects were randomized to treatment: 25 to doxercalciferol and 22 to cholecalciferol.
  Participants
    Female | 9 | 12 | 21
    Male | 16 | 10 | 26
Region of Enrollment [Number; unit: participants]
  United States | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in PTH
Description: Percent reduction in PTH from baseline to 3 months
Time Frame: 3 month
Population: The initial sample size was based on the published response to doxercalciferol versus placebo where a 46% reduction in PTH was observed over 6 months, with a 51% SD. The expected reduction in PTH with cholecalciferol was based on the best-case scenario decrease of 17.8% in PTH with ergocalciferol from our own clinic setting.
Measure: Mean (Standard Deviation); unit: % change in PTH baseline to 3 months
Arm/Group | Doxercalciferol, Active Vitamin D | Cholecalciferol, Inactive Vitamin D
Number analyzed (Participants) | 25 | 22
% change in PTH baseline to 3 months | 27 (34) | 10 (31)

2. Secondary Outcome: Systolic Blood Pressure at 3 Months
Description: systolic blood pressure at 3 months
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Doxercalciferol, Active Vitamin D | Cholecalciferol, Inactive Vitamin D
Number analyzed (Participants) | 25 | 22
mmHg | 120 (47) | 128 (33)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Doxercalciferol, Active Vitamin D | Cholecalciferol, Inactive Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22
Other Adverse Events (participants affected / at risk) | 0/25 | 0/22

LIMITATIONS AND CAVEATS:
Larger, long term studies are needed to demonstrate efficacy of mineral-related and non-mineral-related endpoints and safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No